CLINICAL TRIAL: NCT06681038
Title: Systemic Antitumor Treatment with or Without Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) for Colon Peritoneal Metastases - a Multicentre Phase II Randomized Trial (PIPOX02)
Brief Title: Systemic Antitumor Treatment with or Without Pressurized Intraperitoneal Aerosol Chemotherapy for Colon Peritoneal Metastases (PIPOX02)
Acronym: PIPOX02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2023-14
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Peritoneal Metastases from Colorectal Cancer
Keywords: Surgical oncology; Peritoneal metastasis; Pressurized IntraPeritoneal Aerosol Chemotherapy; Systemic chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control ARM (Active Comparator): Systemic treatments
  Interventions: Drug: Standard Medical Therapy
- Experimental ARM (Experimental): PIPAC procedure with pressurized aerosol containing oxaliplatin.
  Interventions: Drug: Standard Medical Therapy; Procedure: PIPAC

INTERVENTIONS:
Drug: Standard Medical Therapy — Intravenous doublet chemotherapy FOLFIRI or FOLFIRINOX + targeted systemic therapy (anti-EGFR or anti-VEGF).
  Administered every 2 weeks for 12 cycles. Dosage and administration at recommended doses.
Procedure: PIPAC — In addition to standard systemic treatment, patients receive also four PIPAC procedures with pressurized aerosol containing oxaliplatin.
  The PIPAC procedure is repeated up to a maximum of 4 times every 6 weeks.
  Arms: Experimental ARM

SUMMARY:
The goal of this clinical trial is to learn if Pressurized intraperitoneal aerosol chemotherapy (PIPAC) significantly improve the progression-free survival (PFS) in patients with advanced peritoneal metastasis from colorectal cancer.

Researchers will compare 2 strategies, systemic treatments (chemotherapy + targeted therapy) corresponding to standard treatment with or without intraperitoneal oxaliplatin (PIPAC) to see if PIPAC improve the progression-free survival.

Participants will:

* receive a standard treatment every 2 weeks for 12 cycles of intravenous FOLFIRI or FOLFIRINOX + targeted systemic therapy (anti-EGFR or anti-VEGF) in the both arms.
* receive up to a maximum of 4 PIPAC every 6 weeks with pressurized aerosol containing oxaliplatin in experimental arm.
* receive a maintenance treatment until progression or until the onset of severe toxicity after 12 cycles.
* be asked to perform a CT scan and carcinoembryonic antigen (CEA) assay every 8 weeks until progression

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 to 2;
* Histopathologically confirmed colonic adenocarcinoma with synchronous or metachronous peritoneal metastasis (PM);
* Unresectable PM defined as any of the following:

  * PCI >15
  * Extended small bowell involvement
  * Poor general condition contra-indication to a major abdominal surgery (eg: a complete cytoreductive surgery), as decided by the medico-surgical team of the investigator's site specialised in peritoneal carcinomatosis in charge of the patient.
* A surgical exploration performed less than 4 weeks before inclusion (if not, a laparoscopic exploration must be performed);
* First line systemic chemotherapy for advanced / metastatic colonic adenocarcinoma. Systemic chemotherapy in an adjuvant setting is allowed if completed more than 6 months before recurrence and without persistent oxaliplatin-induced neuropathy;
* No extended intraperitoneal adherences defined by at least 9 out of 13 abdominal regions correctly explored during surgical exploration (laparoscopy or laparotomy;

Exclusion Criteria:

* Other cancer treated within the last 3 years, with the exception of in situ cervical carcinoma or basocellular carcinoma;
* Rectal cancer primary (tumor <15 cm from the anal verge);
* Mutational status corresponding to microsatellite instability high (MSI-H) or mismatch repair deficient (dMMR);
* Complete or partial bowel obstruction unresponsive to medical treatment;
* Extraperitoneal polymetastatic diseases. (Only oligometastatic1 diseases are allowed for inclusion);
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess within 6 months prior to enrolment;
* Active gastrointestinal bleeding;
* Inflammatory bowel disease;
* Peripheral neuropathy according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0, grade ≥2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) between the two groups | From randomisation to 18 months after last patient randomisation
  Progression free survival (PFS) is defined as the time (in months) from randomisation until the date of progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) between the two groups | From randomisation to 18 months after last patient randomisation
  Overall survival (OS) defined as the time between randomisation and death from any cause
EORTC QLQ-C30 questionnaire | At enrollment, week 16 and week 32 after the start of treatment
  Quality of life between the two groups evaluated by the score of EORTC QLQ-C30 questionnaire
EORTC QLQ-CR29 questionnaire | At enrollment, week 16 and week 32 after the start of treatment
  Quality of life between the two groups evaluated by the scores of EORTC QLQ-CR29 questionnaire
Peritoneal progression free survival (PPFS) between the two groups | From randomisation to 18 months after last patient randomisation
  Peritoneal progression free survival defined as the time between the date of randomisation and the date of peritoneal progression or death from any cause.
Obstruction-free survival (OFS) between the two groups | From randomisation to 18 months after last patient randomisation
  Obstruction-free survival is defined as the time between the date of randomisation and the appearance of gastrointestinal obstruction requiring medication with high dose of corticosteroïd (> 1mg/kg) or intervention as nasogastric decompression, intraluminal stenting, surgical bypass, or decompression stomy (gastrostomy or ileo/colostomy) or death.
Histological tumor response | At the end of the 12th course of treatment (week 24)
  Peritoneal regression grading score (PRGS) on biopsies performed at surgical exploration in both groups, and systematically during 1st and 2nd PIPAC procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DUMONT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (15):
- France (15):
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - CHU, Lille
  - CHU Dupuytren, Limoges
  - APHM La Timone, Marseille
  - Institut de Cancérologie de Montpellier (ICM), Montpellier
  - APHP Saint Louis, Paris
  - APHP Hôpital Européen Georges Pompidou, Paris
  - Hospices Civils de Lyon - Hôpital Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie de l'Ouest - Saint Herblain, Saint-Herblain
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - CHRU, Strasbourg
  - Centre Hospitalier TARBES, Tarbes
  - Institut de Cancérologie de Lorraine (ICL), Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif